CLINICAL TRIAL: NCT07249151
Title: A Prospective Observational Study Of Early Warning Score Combined With Bedside Assessments In Accelerating Emergency Care Initiation And Improving Patient Prognosis In The Emergency Department
Brief Title: Early Warning Score Combined With Bedside Assessments: Accelerating Emergency Care To Improve Prognosis
Acronym: EWS-BA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jun Liu (Other)
Responsible Party: Sponsor-Investigator, Jun Liu, Attending Physician, Affiliated Hospital of Jiangnan University
Organization: Affiliated Hospital of Jiangnan University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: AHJN-NURS-20240917; 82302187 (Other Grant/Funding Number: National Natural Science Foundation of China)
Record Dates: First submitted 2025-09-17; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Acute Critical Illnesses in Emergency Settings; Process Optimization of Early Warning &Amp; Assessment for At-risk Emergency Patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Optimized ED Bedside Nursing Protocol (Experimental): Arm 1 (Intervention: Optimized ED Assessment) 12 clusters (3 hospitals × 6 depts, day/night shifts) randomized to intervention in 10 phases. Participants get "mNEWS + structured bedside rapid assessment" at triage: 3-min standard assessment (2-min checks: BP, HR, RR, SpO₂, GCS, respiratory status; 1-min mNEWS for risk stratification). Staff prioritize treatment via results. Optimized protocol replaces conventional post-randomization.
  Interventions: Procedure: Optimized ED Bedside Nursing Protocol
- Control Arm: Conventional Emergency Assessment (No Intervention): Control: Conventional ED Assessment Waitlist clusters keep routine assessment pre-randomization. Conventional process: vital sign recording (BP, HR, RR) + subjective severity judgment, no structured scoring/risk stratification. Clusters switch to optimized post-wait, but control data collected only during conventional implementation.

INTERVENTIONS:
Procedure: Optimized ED Bedside Nursing Protocol — A 3-minute standardized emergency nursing assessment exclusively performed by frontline ED nurses, integrating modified National Early Warning Score (mNEWS) and structured bedside checks. Implemented immediately after patient admission (pre-treatment initiation), it includes 2-minute evaluations of systolic BP, HR, RR, SpO₂, respiratory status, and GCS score, followed by 1-minute mNEWS calculation to stratify into low/medium/high risk-directly guiding care prioritization. Distinct from unstructured experience-based assessments or physician-led scoring tools, it's tailored for 24/7 shift-based cluster settings across multiple hospitals.
  Arms: Optimized ED Bedside Nursing Protocol

SUMMARY:
Brief Summary This study, sponsored by the National Natural Science Foundation of China and conducted at the Emergency Department (ED) of Jiangnan University Affiliated Hospital, aims to optimize emergency care for critically ill patients via combining "early warning scoring" and "bedside rapid assessment".

Why the Study? Delayed identification of emergency patients at high risk of deterioration worsens outcomes; traditional assessments often miss subtle deterioration signs. This study seeks a more efficient assessment approach to help clinicians recognize high-risk patients earlier and start targeted treatment faster.

Eligibility 200-300 participants will be recruited from the hospital's ED for acute diseases (e.g., severe infection, heart failure, trauma). Inclusion: aged 18-80, with informed consent (or family consent if unable to communicate). Exclusion: severe mental illness, non-intervenable terminal illness.

Study Process All participants receive routine emergency care. The research team uses a new combined assessment tool: first a 2-minute bedside rapid assessment (vital signs, consciousness, breathing), then early warning scoring to classify risk. Doctors adjust treatment priority based on results. The team records time from admission to treatment initiation and 72-hour condition changes. No additional invasive procedures/experimental drugs are used, and no extra cost for assessments.

Potential Benefits Participants may get more timely, targeted emergency care (reducing deterioration risk and hospital stay). Study results will improve emergency care at this and other hospitals, benefiting more emergency patients.

Study Leadership Principal Investigator: Dr. Jun Liu (Attending Physician, ED of Jiangnan University Affiliated Hospital) Responsible Party: Jiangnan University Affiliated Hospital (Sponsor) Ethical Approval: Approved by the hospital's Medical Ethics Committee (Approval No.: To be filled with actual number)

ELIGIBILITY:
Inclusion Criteria:

Patients will be eligible for enrollment if they meet all of the following conditions:

1. Age between 18 and 80 years at the time of presentation.
2. Presentation to the emergency department (ED) for acute medical evaluation.
3. Completion of at least one documented Early Warning Score (EWS) assessment upon ED admission or during the ED stay.

Exclusion Criteria:

Patients will be excluded if they meet any of the following criteria:

1. Do-not-resuscitate (DNR) orders or enrollment in a palliative/comfort care pathway at the time of presentation.
2. Cardiac arrest upon arrival to the ED (unresponsive, pulseless, requiring resuscitation without return of spontaneous circulation).
3. Transfer out of the hospital (to another institution or to the operating room for immediate surgery) within 24 hours of ED admission.
4. History of major cardiac surgery (e.g., coronary artery bypass grafting, valve replacement) or heart transplantation, as these conditions may alter baseline hemodynamics and limit EWS applicability.
5. Severe chronic organ dysfunction, including:

   End-stage renal disease requiring maintenance dialysis; Severe hepatic insufficiency (Child-Pugh class C or equivalent); Advanced heart failure (New York Heart Association class IV).
6. Known allergy or contraindication to iodinated contrast media (if relevant laboratory or imaging assessments are required for outcome evaluation).
7. Pregnancy, due to altered physiological parameters and ethical considerations.
8. Incomplete or missing clinical records, preventing calculation of EWS or confirmation of study endpoints.
9. Duplicate enrollment due to repeated ED visits or readmissions during the study period (only the first eligible admission will be included).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-08-30 (Actual); Study Completion 2025-09-16 (Actual)

PRIMARY OUTCOMES:
ICU-Level Organ Support or In-Hospital Mortality Within 24 Hours | From the time of patient admission (admission time) up to 24 hours after admission time.
  Composite endpoint defined as the occurrence of either "ICU-level organ support" or "in-hospital mortality" within 24 hours after EWS score ≥5 (T0). "ICU-level organ support" includes: invasive mechanical ventilation initiation, continuous vasopressor use for ≥30 minutes, or CRRT activation. "In-hospital mortality" refers to death occurring during the current hospitalization. Data are extracted from electronic medical records (EMR) and ICU information systems, with event time confirmed by the earliest timestamp of organ support initiation or death notification.

SECONDARY OUTCOMES:
T3 Compliance Rate | Within the first 24 hours from ED registration
  T3 is a time-limited indicator for the process "Junior Nurse (JN) reporting → Senior Nurse (SN) secondary assessment". The time frame focuses on the maximum observation window (≤10 minutes) of this process, directly linking to the "time limit criteria" for compliance rate.
Door-to-Key Intervention Time | Within the first 24 hours from ED registration
  The core of "door-to-intervention time" is the interval between "registration time → intervention execution time". The time frame covers the complete timing cycle, adapting to the phenotype-stratified intervention logic.intervention execution time". The time frame covers the complete timing cycle, adapting to the phenotype-stratified intervention logic.
72-Hour ICU Admission Rate | From T0 (time of enrollment or index event) until ICU admission or hospital discharge, whichever occurs first, assessed up to 72 hours post-T0.
  This outcome measure focuses on the rate of ICU admission within the "72-hour post-T0" window. Observation terminates if the patient is discharged from the hospital before 72 hours post-T0 (and no ICU admission occurs during the hospitalization). The unit of measure is a percentage (%).
28-Day In-Hospital Mortality | From patient ED registration up to 28 days after registration
  This outcome measure focuses on in-hospital mortality within the "28-day post-registration" window. Observation terminates at the earlier of two events: ① the patient's death during hospitalization, or ② the patient's discharge from the hospital (if no death occurs during the 28-day post-registration period). The unit of measure is a percentage (%).
Incidence of Over-Escalation and Delayed Escalation | From T0 (initial escalation decision) until confirmation of intervention necessity or time limit deviation, whichever occurs first, assessed up to 72 hours post-T0.
  Over-escalation requires a "72-hour observation period to verify intervention necessity", while delayed escalation requires immediate determination of time limit deviation. The time frame aligns with the judgment logic of both events.

CONTACTS AND LOCATIONS:
Locations (1):
- Wuxi Taihu Hospital; Affiliated Hospital of Jiangnan University; Wuxi Binhu District Traditional Chinese Medicine Hospital; Wuxi Xinwu District Traditional Chinese Medicine Hospital, Wuxi, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data (IPD) are pending final quality inspection, consistency verification, and standardized organization; premature sharing may lead to the use of unvalidated data, thereby compromising the reliability of secondary analyses. The current IPD will support subsequent sub-studies (e.g., disease phenotype-stratified analysis, long-term outcome correlation research). Temporary non-sharing of data prevents the redundant use of core data and ensures the integrity of this research series.
  Upon completion of the aforementioned tasks (final data verification, implementation of follow-up sub-studies, confirmation of data security), the team will re-evaluate the IPD sharing arrangement. If feasible, the relevant arrangements will be promptly disclosed via ClinicalTrials.gov.

REFERENCES:
- [Result] Covino M, Sandroni C, Della Polla D, De Matteis G, Piccioni A, De Vita A, Russo A, Salini S, Carbone L, Petrucci M, Pennisi M, Gasbarrini A, Franceschi F. Predicting ICU admission and death in the Emergency Department: A comparison of six early warning scores. Resuscitation. 2023 Sep;190:109876. doi: 10.1016/j.resuscitation.2023.109876. Epub 2023 Jun 17. PMID 37331563
- [Result] Churpek MM, Snyder A, Han X, Sokol S, Pettit N, Howell MD, Edelson DP. Quick Sepsis-related Organ Failure Assessment, Systemic Inflammatory Response Syndrome, and Early Warning Scores for Detecting Clinical Deterioration in Infected Patients outside the Intensive Care Unit. Am J Respir Crit Care Med. 2017 Apr 1;195(7):906-911. doi: 10.1164/rccm.201604-0854OC. PMID 27649072
- [Result] Candel BGJ, Nissen SK, Nickel CH, Raven W, Thijssen W, Gaakeer MI, Lassen AT, Brabrand M, Steyerberg EW, de Jonge E, de Groot B. Development and External Validation of the International Early Warning Score for Improved Age- and Sex-Adjusted In-Hospital Mortality Prediction in the Emergency Department. Crit Care Med. 2023 Jul 1;51(7):881-891. doi: 10.1097/CCM.0000000000005842. Epub 2023 Mar 23. PMID 36951452
- [Result] Arevalo-Buitrago P, Morales-Cane I, Olivares Luque E, Godino-Rubio M, Rodriguez-Borrego MA, Lopez-Soto PJ. Early detection of risk for clinical deterioration in emergency department patients: validation of a version of the National Early Warning Score 2 for use in Spain. Emergencias. 2022 Dec;34(6):452-457. English, Spanish. PMID 36625695
- [Result] Nannan Panday RS, Minderhoud TC, Alam N, Nanayakkara PWB. Prognostic value of early warning scores in the emergency department (ED) and acute medical unit (AMU): A narrative review. Eur J Intern Med. 2017 Nov;45:20-31. doi: 10.1016/j.ejim.2017.09.027. Epub 2017 Oct 7. PMID 28993097